CLINICAL TRIAL: NCT07359456
Title: Randomized Phase 2 Study of Second-line Chemotherapy Comparing FOLFIRI + Ivonescimab Versus FOLFIRI + Bevacizumab in Microsatellite Stable (MSS)/ Proficient MisMatch Repair (pMMR) BRAF Wild Type (BRAFwt) Advanced Colorectal Cancer (mCRC) Without Liver Metastases
Brief Title: Testing Ivonescimab in Combination With Chemotherapy in Patients With Metastatic Colorectal Cancers Without Liver Metastases
Acronym: COLIBRI-GI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-GIG-2518; 2025-524215-36-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-09; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; ivonescimab; BRAF wild-type
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivonescimab + FOLFIRI (Experimental): Ivonescimab 20 mg/kg by intravenous infusion (IV) once every 2 weeks (Q2W) combined with FOLFIRI chemotherapy (irinotecan 180 mg/m2 IV, folinic acid 400 mg/m2 IV (or L-folinic acid 200 mg/m²), and fluorouracil (5-FU) 400 mg/m² IV bolus; followed by 5 FU 2400 mg/m2 as a 46 hour continuous IV infusion), every two weeks
  Interventions: Drug: Ivonescimab; Drug: FOLFIRI Protocol
- Bevacizumab + FOLFIRI (Active Comparator): Bevacizumab 5 mg/kg by intravenous infusion (IV) once every 2 weeks (Q2W) combined with FOLFIRI chemotherapy (irinotecan 180 mg/m2 IV, folinic acid 400 mg/m2 IV (or L-folinic acid 200 mg/m²), and fluorouracil (5-FU) 400 mg/m² IV bolus; followed by 5 FU 2400 mg/m2 as a 46 hour continuous IV infusion), every two weeks
  Interventions: Drug: Bevacizumab; Drug: FOLFIRI Protocol

INTERVENTIONS:
Drug: Ivonescimab — Ivonescimab 20 mg/kg by intravenous infusion (IV) once every 2 weeks (Q2W)
  Arms: Ivonescimab + FOLFIRI
Drug: Bevacizumab — Bevacizumab 5 mg/kg by intravenous infusion (IV) once every 2 weeks (Q2W)
  Arms: Bevacizumab + FOLFIRI
Drug: FOLFIRI Protocol — FOLFIRI chemotherapy (irinotecan 180 mg/m2 IV, folinic acid 400 mg/m2 IV (or L-folinic acid 200 mg/m²), and fluorouracil (5-FU) 400 mg/m² IV bolus; followed by 5 FU 2400 mg/m2 as a 46 hour continuous IV infusion), every two weeks

SUMMARY:
The goal of this clinical trial is to evaluate the superiority of ivonescimab combined with FOLFIRI over FOLFIRI + bevacizumab as second-line treatment of non resectable pMMR/MSS BRAFwt mCRC patients without liver metastases in terms of PFS. The main questions it aims to answer are:

Does FOLFIRI + ivonescimab improve progression-free survival compared to FOLFIRI + bevacizumab?

Participants will:

Take FOLFIRI + ivonescimab or FOLFIRI + bevacizumab every 2 weeks for a maximum of 24 months Visit the clinic once every 2 weeks for checkups and tests, and have imaging done every 8 weeks Complete some quality of life questionnaires every 8 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Signed a written informed consent form prior to any trial specific procedures. Note: If the patient is physically unable to provide their written consent, a trusted person of their choice, independent of the Investigator or the Sponsor, can confirm the patients consent in writing.
2. Histologically confirmed diagnosis of non resectable pMMR (by IHC) and MSS (by molecular biology) and BRAFwt metastatic colorectal cancer with no liver metastasis.
3. Must have previously received 1st-line treatment with FOLFOX +/- anti-VEGF (Vascular endothelial growth factor) or EGFR (Epithelial Growth Factor Receptor) therapy (including recurrence within 6 months after adjuvant FOLFOX for localized CRC and adjuvant/perioperative FOLFOX for mCRC, as well as progressive disease under maintenance treatment for mCRC) OR 1st-line treatment with FOLFIRINOX (Oxaliplatin, Irinotecan, 5FU, Folinic acid) (under the following condition: no progression under triplet-chemotherapy, progression under LV5FU2 (Folinic acid + 5FU) maintenance, irinotecan stopped for at least 3 months for a reason other than progression)
4. Presence of at least one measurable lesion as assessed by the investigator according to RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Age ≥18 years.
7. Adequate Organ Function:

   * Hematology (no blood transfusions or growth factor therapy used within 7 days of the screening):

     * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
     * Platelet count ≥ 100 × 109/L
     * Hemoglobin ≥ 10.0 g/dL
   * Kidneys:

     * Creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault formula or estimated glomerular filtration rate (eGFR) value ≥50 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
     * Urine protein < 2+ or 24 hour urine protein quantification < 1.0 g
   * Liver:

     * Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN)
     * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN
   * Coagulation: prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5 x ULN, and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN (unless abnormalities are unrelated to coagulopathy, or prophylactic coagulation)
8. Life expectancy ≥ 3 months
9. Women of childbearing potential (WOCBP) having sex with an unsterilized male partner and unsterilized males having sex with a female partner of childbearing potential, must agree to use an effective method of contraception for the duration of trial participation and as required after completing study treatment (9 months after the last dose of trial treatment). Men must also agree to not donate sperm and women must agree to not donate oocytes during the specified period.
10. WOCBP must have a negative serum pregnancy test performed within 3 days before inclusion and a negative urine pregnancy test on the day of first dose, prior to treatment administration.
11. Willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests, and other study procedures
12. Affiliation to the Social Security System (or equivalent)

Exclusion Criteria:

1. Presence of liver metastases by CT-scan or MRI. Note: Patients with prior definitively treated liver metastases (surgical resection, microwave or radiofrequency ablation, or stereotactic body radiation therapy) are eligible if no evidence of metastatic disease in the liver on subsequent imaging).
2. History of Gilbert's syndrome
3. Other current or previous malignancy within the past 3 years (with the exception of squamous cell carcinoma of the skin or in situ tumour treated by surgery).
4. Patients with high microsatellite instability (MSI-H), mismatched repair disease (dMMR) and/or BRAF V600E mutated tumor.
5. Toxicities from previous treatment not resolved to grade ≤ 1 (according to the version 5.0 of the National Cancer Institute - Common terminology criteria for adverse events [NCI-CTCAE v5.0]) before treatment start with the exception of alopecia.
6. Major surgical procedures or serious trauma within 4 weeks prior to randomization, or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to randomization.
7. History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to randomization, including but not limited to:

   * Clinically significant GI bleeding such as hematochezia or any episodes of melena or documented acute hemoglobin drop of more than 1 gm in 2 weeks prior to randomization
   * Current use of prophylactic or full-dose anticoagulants or anti-platelet agents for therapeutic purposes that is not stable prior to randomization is not allowed. The use of full-dose anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits according to the medical standard of the enrolling institution.
8. Current hypertension with systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy
9. History of major diseases before randomization, specifically:

   * Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association (NYHA) classification ≥ grade 2) or vascular disease (eg, aortic aneurysm at risk of rupture) that required hospitalization within 12 months prior to randomization, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia)
   * History of oesophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months before randomization
   * History of arterial thromboembolic event, venous thromboembolic event of Grade 3 and above as specified in National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to randomization
   * Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks before randomization
   * History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to randomization
10. Current presence of significant radiographic or clinical manifestations of gastrointestinal (GI) obstruction.
11. Ascites requiring paracentesis within last 30 days
12. Symptomatic central nervous system (CNS) metastases or leptomeningeal disease Note: Asymptomatic patients (previously treated or untreated) in the absence of corticosteroid and anti-epileptic therapy are allowed. CNS metastases must be stable for ≥4 weeks prior to randomization.
13. Presence of brainstem, meningeal metastases, spinal cord metastases, or compression.
14. Active or prior history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea)
15. Prior immunosuppressive therapy: immunosuppressive doses of systemic medications of > 10 mg/day of prednisone or equivalent must be discontinued ≥ 2 weeks before the first dose of study treatment. Short courses of high dose corticosteroids and/or continuous low dose of prednisone (< 10 mg/day) are permitted. In addition, inhaled, intranasal, intraocular, and/or joint injections of corticosteroids are allowed.
16. Any prior clinically significant or active autoimmune disease requiring systemic therapy (eg, with disease- modifying drugs, prednisone >10 mg daily or equivalent, immunosuppressant therapy or immunomodulatory agents [eg, infliximab or IVIG (intravenous immunoglobulin)]) within 2 years prior to randomization; however, the following will be allowed:

    o Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is permitted.
17. Known history of, or any evidence of, interstitial lung disease.
18. Patient with non-controlled human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) infection (patient with undetectable viral load (HIV RNA PCR) and CD4 (T CD4 lymphocytes) above 350 either spontaneously or on stable anti-viral regimen).
19. Known human immunodeficiency virus infection with CD4+ T cell counts < 350 cells/µL, hepatitis C infection (subjects with hepatitis C who achieve a sustained virologic response following antiviral therapy are permitted), or hepatitis B infection (subjects with hepatitis B surface antigen or core antibody who achieve sustained virologic response with antiviral therapy directed at hepatitis B are permitted)
20. Proven complete deficiency of dihydropyrimidine dehydrogenase (DPD).
21. Known history of hypersensitivity to ivonescimab and to one of the study drugs or one of its excipients
22. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol.
23. Pregnant or breast-feeding females.
24. Participation in another therapeutic trial within the 30 days prior to entering the study. Participation in an observational trial would be acceptable.
25. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons.
26. Individuals deprived of liberty or placed under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Time from the date of randomization until the date of first documented disease progression as assessed by the investigator according to RECIST1.1, or death from any cause, whichever came first, assessed up to 72 months.
  The primary objective is to evaluate the superiority of ivonescimab combined with FOLFIRI over FOLFIRI + bevacizumab as second-line treatment of non resectable pMMR/MSS BRAFwt mCRC patients without liver metastases in terms of Progression-Free Survival (PFS).

SECONDARY OUTCOMES:
PFS as per iRECIST | The time from the date of randomization to the date of first documentation of disease progression as assessed by the investigator according to iRECIST, or death from any cause, whichever came first, assessed up to 72 months.
  To evaluate the efficacy of ivonescimab in combination with FOLFIRI in terms of PFS as per iRECIST
Overall Response Rate (ORR) as per RECIST v1.1 | Imagery will be done within 28 days before first study treatment, and every 8 weeks until the date of the first documented disease progression.
  To evaluate the efficacy of ivonescimab in combination with FOLFIRI in terms of Overall Response Rate (ORR) as per RECIST v1.1. The proportion of patients achieving complete response (CR) or partial response (PR) as assessed by the investigator according to RECIST v1.1.
Duration of Response (DOR) as per RECIST v1.1 | The time from first documented PR or CR (compared to baseline measurement done within 28 days before first study treatment) until the date of PD (Imagery done every 8 weeks), or death from any cause.
  To evaluate the efficacy of ivonescimab in combination with FOLFIRI in terms of Duration of Response (DOR) as per RECIST v1.1.
Overall Survival (OS) | From date of randomization until the date of death from any cause, whichever came first, assessed up to 72 months.
  To evaluate the efficacy of ivonescimab in combination with FOLFIRI in terms of Overall Survival (OS). The time from randomization to death from any cause. Patients who are alive at the data-cutoff date will be censored on the last known alive date.
Safety and tolerability of treatment (NCI-CTCAE version 5.0) | At baseline within 14 days prior first study treatment, at day 1 of each visit during treatment (every 2 weeks), at the end of treatment (30 days after last study treatment), and at the two first follow-up (every 8 weeks after last administration).
  Toxicity / Adverse events (AEs), occurrence of treatment-related AEs, treatment-related AEs (TRAEs) leading to dose reduction or discontinuation during treatment, serious adverse events (SAEs) and suspected unexpected serious adverse reactions (SUSARs), iand tolerability of treatment (NCI-CTCAE version 5.0)
The effect of treatments on Quality of Life (QoL) - QLQ-C30 | At baseline within 14 days prior first study treatment, every 8 weeks from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 72 months
  QoL is assessed using the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaires QLQ-C30 and EORTC QLQ-CR29
The effect of treatments on Quality of Life (QoL) - QLQ-CR29 | At baseline within 14 days prior first study treatment, every 8 weeks from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 72 months
  QoL is assessed using the European Organisation for Research and Treatment of Cancer

CONTACTS AND LOCATIONS:
Locations (22):
- France (22):
  - CH d'Auxerre, Auxerre
  - Centre Hospitalier de Beuvry, Beuvry
  - Centre François Baclesse, Caen
  - CH de Calais, Calais
  - Polyclinique Saint Côme, Compiègne
  - Institut Andrée Dutreix, Coudekerque-Branche
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Européen de Marseille, Marseille
  - Hôpital la Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - CHRU de Nancy, Nancy
  - Hôpital Saint Antoine - APHP, Paris
  - Hôpital Saint Louis - APHP, Paris
  - Hôpital Privé des côtes d'Armor, Plérin
  - CHU de Poitiers, Poitiers
  - CHU de Reims, Reims
  - Institut Jean Godinot, Reims
  - CHU de Rouen, Rouen
  - Institut de Cancérologie de l'Ouest - Site René Gauducheau, Saint-Herblain
  - Centre Hospitalier de Valenciennes, Valenciennes
  - Gustave Roussy, Villejuif